CLINICAL TRIAL: NCT01592617
Title: Phase II Study of Peptide Cancer Vaccine S-488410 to Treat Advanced Non-Small Cell Lung Cancer
Brief Title: Phase II Study of S-488410 to Treat Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shiga University (Other)
Collaborators: Showa University (Other); Fukushima Medical University (Other); Tohoku University (Other); Shionogi (Industry); Tokyo University (Other); University of Chicago (Other)
Responsible Party: Principal Investigator, Yataro Daigo, Professor of Medical Oncology, Director of Cancer Center, Shiga University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S488410LP; UMIN000007873 (Registry Identifier: UMIN: University Hospital Medical Information Network)
Record Dates: First submitted 2012-05-02; First posted 2012-05-07 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: cancer vaccine; HLA-A*24:02; lung cancer; CTL
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- S-488410 (Experimental)
  Interventions: Drug: S-488410

INTERVENTIONS:
Drug: S-488410 — In multicenter HLA-blinded open study, patients will be vaccinated subcutaneously once a week with S-488410 (S-488401, S-488402, S-488403, 1mg each).
  Other Names: S-488410 (S-488401, S-488402, S-488403).

SUMMARY:
The investigators identified three cancer-testis antigens, as targets for cancer vaccination against lung cancer. In this clinical study, the investigators examine using a combination of three peptides from these three antigens (S-488410) the safety, immunogenicity, and antitumor effect of vaccine treatment for advanced non-small cell lung cancer patients.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the clinical efficacy and safety of S-488410 for advanced non-small cell lung cancers who failed to standard therapy.

The investigators previously identified three novel HLA-A*2402-restricted epitope peptides, which were derived from three cancer-testis antigens, as targets for cancer vaccination against lung cancer. In this phase II trial, we examine using a combination of these three peptides the safety, immunogenicity, and antitumor effect of vaccine treatment for HLA-A*2402-positive advanced small cell lung cancer patients who failed to standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Advanced NSCLC that cannot undergo curative surgery.
* Patients that are refractory to standard chemotherapy or cannot be treated with further therapy due to severe adverse effects of chemotherapy.
* Histologically diagnosed NSCLC.
* Clinical efficacy can be evaluated by radiologic methods within 4 weeks prior to receiving treatment.
* ECOG performance status 0-2 within 2 weeks prior to receiving treatment.
* Life expectancy > 3 months.
* Age between 20 to 79
* Male or Female.
* In patients or out patients.
* Able and willing to give valid written informed consent.

Exclusion Criteria:

* Other malignancy requiring treatment
* radiation, immunotherapy, hyperthermia, or surgery.
* Active and uncontrolled infectious disease
* Active and uncontrolled hepatic dysfunction, kidney dysfunction, cardiac disease, or lung disease (i.e. interstitial pneumonia).
* Autoimmune disease.
* HIV-Ab or antigen positive
* Prior anti-cancer therapy within 4 weeks
* Laboratory values as follows: 2000<mm3 < WBC < 15000/mm3, Platelet count < 50000/mm3, Asparate transaminase > 5 X cutoff value, Alanine transaminase > 5 X cutoff value, Total bilirubin > 3 X cutoff value, and Serum creatinine > 3X cutoff value.
* Patients knows HLA-A type.
* Breastfeeding and Pregnancy (woman of child bearing potential)
* Refusal of pregnancy conception.
* Treated with S-488401, S-488402, or S-488403.
* Treated with other investigational drug within 3 months prior to receiving S-48810 treatment.
* Decision of nonenrollment of the patients by principal investigator or physician-in-charge from the view point of patient's safety.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2012-05; Primary Completion 2015-08 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Evaluation of difference in overall survival after vaccination therapy between HLA-A 24:02 and non-HLA-A 24:02 patients. | Participants will be followed for the duration of vaccination therapy, an expected average of more than 1 year.

SECONDARY OUTCOMES:
CTL response between HLA-A24:02 and non-HLA-A24:02 | Participants will be followed for the duration of vaccination therapy, an expected average of more than 1 year.
PFS and ORR between HLA-A24:02 and non-HLA-A24:02 | Participants will be followed for the duration of vaccination therapy, an expected average of more than 1 year.
PFS and OS between CTL response positive and negative | Participants will be followed for the duration of vaccination therapy, an expected average of more than 1 year.
Safety and tolerability: Number of Adverse Events with information of disease, grade and incidence | Participants will be followed for the duration of vaccination therapy, an expected average of more than 1 year.
Identification of biomarkers for efficacy and safety that are mentioned above | Participants will be followed for the duration of vaccination therapy, an expected average of more than 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Yataro Daigo, MD, PhD, Principal Investigator — Department of Medical Oncology, Shiga University of Medical Science
Locations (1):
- Department of Medical Oncology, Shiga University of Medical Science Hospital, Ōtsu, Shiga, Japan

REFERENCES:
- [Background] Kono K, Mizukami Y, Daigo Y, Takano A, Masuda K, Yoshida K, Tsunoda T, Kawaguchi Y, Nakamura Y, Fujii H. Vaccination with multiple peptides derived from novel cancer-testis antigens can induce specific T-cell responses and clinical responses in advanced esophageal cancer. Cancer Sci. 2009 Aug;100(8):1502-9. doi: 10.1111/j.1349-7006.2009.01200.x. Epub 2009 May 14. PMID 19459850
- [Background] Harao M, Hirata S, Irie A, Senju S, Nakatsura T, Komori H, Ikuta Y, Yokomine K, Imai K, Inoue M, Harada K, Mori T, Tsunoda T, Nakatsuru S, Daigo Y, Nomori H, Nakamura Y, Baba H, Nishimura Y. HLA-A2-restricted CTL epitopes of a novel lung cancer-associated cancer testis antigen, cell division cycle associated 1, can induce tumor-reactive CTL. Int J Cancer. 2008 Dec 1;123(11):2616-25. doi: 10.1002/ijc.23823. PMID 18770861
- [Background] Mizukami Y, Kono K, Daigo Y, Takano A, Tsunoda T, Kawaguchi Y, Nakamura Y, Fujii H. Detection of novel cancer-testis antigen-specific T-cell responses in TIL, regional lymph nodes, and PBL in patients with esophageal squamous cell carcinoma. Cancer Sci. 2008 Jul;99(7):1448-54. doi: 10.1111/j.1349-7006.2008.00844.x. Epub 2008 Apr 30. PMID 18452554
- [Background] Daigo Y, Nakamura Y. From cancer genomics to thoracic oncology: discovery of new biomarkers and therapeutic targets for lung and esophageal carcinoma. Gen Thorac Cardiovasc Surg. 2008 Feb;56(2):43-53. doi: 10.1007/s11748-007-0211-x. Epub 2008 Feb 24. PMID 18297458
- [Background] Ishikawa N, Takano A, Yasui W, Inai K, Nishimura H, Ito H, Miyagi Y, Nakayama H, Fujita M, Hosokawa M, Tsuchiya E, Kohno N, Nakamura Y, Daigo Y. Cancer-testis antigen lymphocyte antigen 6 complex locus K is a serologic biomarker and a therapeutic target for lung and esophageal carcinomas. Cancer Res. 2007 Dec 15;67(24):11601-11. doi: 10.1158/0008-5472.CAN-07-3243. PMID 18089789
- [Background] Suda T, Tsunoda T, Daigo Y, Nakamura Y, Tahara H. Identification of human leukocyte antigen-A24-restricted epitope peptides derived from gene products upregulated in lung and esophageal cancers as novel targets for immunotherapy. Cancer Sci. 2007 Nov;98(11):1803-8. doi: 10.1111/j.1349-7006.2007.00603.x. PMID 17784873
- [Background] Hayama S, Daigo Y, Kato T, Ishikawa N, Yamabuki T, Miyamoto M, Ito T, Tsuchiya E, Kondo S, Nakamura Y. Activation of CDCA1-KNTC2, members of centromere protein complex, involved in pulmonary carcinogenesis. Cancer Res. 2006 Nov 1;66(21):10339-48. doi: 10.1158/0008-5472.CAN-06-2137. PMID 17079454